CLINICAL TRIAL: NCT02185157
Title: Effects of Dual-task Versus Aerobic Training on Gait Stride Variability and Cognitive Function of Independent Community-dwelling Elderly Women: A Randomized Controlled Trial
Brief Title: Effects of Dual-task Exercises on Gait Parameters and Cognitive Function in Elderly Women: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Gisele de Cássia Gomes, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECAGGOMESUFMG -001; CAAE 0448.0.203.000-11 (Registry Identifier: Comite de Ética em Pesquisa da UFMG)
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: elderly; dual-task training; aerobic training; gait; cognition
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Dual Task exercises (Experimental): Dual-task training, includes 18 sessions model of cognitive and 12 motor dual-task exercises model, were administered in groups of four participants in a comfortable environment, without distraction effects. The 50-minute sessions included 30 minutes of motor dual-task exercises, and then, the participants were divided into pairs. The first pair performed free walks during 10 minutes at their maximal speeds, while the other received individual cognitive dual-task training for the same time, and these activities will be exchanged, so that all pairs could walk and receive cognitive training.
  Interventions: Other: dual -task exercises
- Control intervention: Aerobic training (Other): The same doses of aerobic training, i.e., 50 minutes, was delivered in groups of five participants. Each session will include 10 minutes of warm-up, 30 minutes of aerobic training on an ergometric bicycle at 60 to 80% of the participants' maximum heart rates,and 10 minutes of cool-down exercises.
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: dual -task exercises — physical exercises sections with gait and a second task like talk answering some questions or making some exercise with the arms.
  Other Names: physical exercises; aerobic training; physical activity
  Arms: Experimental: Dual Task exercises
Other: Aerobic training — The same doses of aerobic training, i.e., 50 minutes, was delivered in groups of five participants. Each session will include 10 minutes of warm-up, 30 minutes of aerobic training on an ergometric bicycle at 60 to 80% of the participants' maximum heart rates,and 10 minutes of cool-down exercises.
  Arms: Control intervention: Aerobic training

SUMMARY:
The training of a secondary task while walking, whether it is reasoning activities, memory or motor tasks, may enhance automation, walking performance, and postural control and, thus, minimize the risk of falls influenced by the walking patterns variability. However, the literature is scarce regarding the influence of dual-task training on changes in gait parameters.

The purpose of this prospective, blinded randomized controlled trial is to compare the short- and long-term effects of dual-task and aerobic training on gait stride variability and superior cerebral functions of independent community-dwelling elderly women.

The participants will be randomly allocated into either experimental or control groups.The experimental group will undertake 50 minutes/day of dual-task training, three times/week over 12 weeks, totaling 36 sessions, whereas the control group will receive the same doses of aerobic training. At baseline, after 18 and 36 sessions, and 12 weeks after the cessation of the interventions, researchers blinded to group allocations will collect the outcome measures.The interventions will be delivered by trained physical therapists.

Primary outcome will include gait stride variability, which will be assessed by a movement analysis system: the GaitRite® system, during cognitive and motor dual-tasks, at both normal and fast speeds. Secondary outcome measures will include a battery of global and specific cognitive function tests.

The findings of this trial may help better understand whether cognitive-motor interventions with older adults, when compared to traditional aerobic training, would result in greater improvements in gait under dual-task conditions and lead to improvements in cognitive tasks. Furthermore, the findings could potentially bring important insights regarding the impacts of improvements in walking abilities and cognition.

DETAILED DESCRIPTION:
Socially speaking, the findings could potentially bring important insights regarding the impacts of improvements in walking abilities and cognition. If the elderly maintain safe gait patterns that prevent falls, they could reach self-sustained community participation and consequently reduce the burden of care on the family and caregivers. Additionally, the public health system may ultimately receive important positive economic and social impacts. This clinical trial may be reproduced in research and clinical practice environments.

ELIGIBILITY:
Inclusion Criteria:

* Elderly women will be eligible if they are between 69 and 79 years of age, have at least three years of schooling,have no cognitive deficits, as determined by the scores on the Mini-Mental State Examination, adjusted for their education levels: ≥23 for three years, ≥25 for four to seven years, and ≥26 for eight or more years of school.

Exclusion Criteria:

* Participants will be excluded if they have neuromusculoskeletal diseases,which could restrain physical activities or make use of medications, which could interfere with motor performance and/or memory.

Ages: 69 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
change of gait stride variability | Baseline, at the sixth week as a intermediary measure, final and three months after the end of the study
  The change in gait stride variability will be measured by a movement analysis system: The GaitRite® system that gives another gait parameters as speed, step width, double support, etc.

SECONDARY OUTCOMES:
Changes on the Executive function measured by Addenbrooke's Cognitive Examination-Revised (ACE-R) | baseline, at the sixth week as a intermediary measure, final and three months after the end of study months later
  This outcome measure will be assessed by the Brazilian version of the Addenbrooke's Cognitive Examination-Revised (ACE-R) that is a global cognitive assessment instrument with high sensitivity and specificity to detect mild dementia and differentiate frontotemporal dementia from Alzheimer's disease. This instrument assess orientation and attention, memory, verbal fluency, language and visual-spatial skills.
  A maximum score of 100 is calculated from five sub-scores: Orientation and attention (18 points); memory (26 points); verbal fluency (14 points); language (26 points); and visual-spatial skills (16 points) [26]. The validation study of the English version of the ACE-R proposed a cut-off score of 88 points for higher sensitivity (sensitivity 94 %, specificity89 %). A cut-off score of 82 points was proposed for better specificity (specificity: 100 %, sensitivity: 84%), with population-based norms also available for the Brazilian population.

OTHER OUTCOMES:
Changes on Stroop test or the Color-word interference test | Baseline,at the sixth week as a intermediary measure, final and three months after the end of the study
  This test consists of two tasks. For the first task, the participants are asked to name, as fast as possible, the color seen in a square with various color circles. Then, the same colors are shown as written words, instead of the circles. However, the colors are printed in an incongruent way, that is, the word is written in red, but the color is yellow and the participant should be able to identify the color, and not read the word. The examiner takes note of the time and the number of mistakes. The Stroop effect is said to be the difference between the time of execution of the first and the second tasks. Both the time, in minutes, and the number of errors will be registered for analyses.
Changes on Trail making test | Baseline, at the sixth week as a intermediary measure, final and three months after the end of the study
  The trail making test is a classic executive function test and several studies have shown the relationships between its scores with gait abilities. Overall, the test assesses the time to execute visual-motor tasks, as a dimension of a cognitive flexibility test.The test includes two parts:The first consists of drawing a simple line that requires that the individual links numbers 1 to 25, consecutively.The second requires the same consecutive number linking, but now have the interference of letters, so that the linkage is made by alternating letters and numbers. It is also a time-measured test and the time, in minutes, to conclude both parts, will be registered for analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Gisele C. Gomes, Master, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Department of Physical Therapy, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- See also: University — http://www.ufmg.br